CLINICAL TRIAL: NCT03795402
Title: Collection of Skin Punch Biopsies and Non-Invasively Collected Microneedle Device Samples From Subjects With Mild Chronic Plaque Psoriasis Vulgaris to Use for Transcriptomics Profiling
Brief Title: Analysis of Non-Invasively Collected Microneedle Device Samples From Mild Plaque Psoriasis for Use in Transcriptomics Profiling
Status: Completed | Type: Observational
Sponsor: Janssen Research & Development, LLC (Industry)
Collaborators: Innovaderm Research Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: 8004053; 8004053 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2019-01-04; First posted 2019-01-07 (Actual); Last update posted 2019-12-13 (Actual); Status verified 2019-12

CONDITIONS: Psoriasis Vulgaris

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A: Three microneedle device samples will be collected from a psoriasis lesion and from nonlesional (healthy) skin on Day 1. Two skin biopsies of 4 millimeter (mm) will be performed on Day 1. No investigational drug product will be administered during this study.
  Interventions: Device: Microneedle Device
- Group B: One microneedle device sample will be collected from a psoriasis lesion and from nonlesional (healthy) skin on Day 1 and at Weeks 2 and 4. Two skin biopsies of 4 mm will be performed on Day 1. No investigational drug product will be administered during this study.
  Interventions: Device: Microneedle Device

INTERVENTIONS:
Device: Microneedle Device — Microneedle device will be used for collecting skin samples as a non-invasive method.

SUMMARY:
The purpose of this study is to collect skin biopsies and non-invasive microneedle device samples from participants with mild chronic plaque psoriasis vulgaris to use for transcriptomics profiling for further investigation.

ELIGIBILITY:
Inclusion Criteria:

* Participant has a history of chronic plaque psoriasis vulgaris for at least 6 months prior to the screening visit
* Participant has had stable psoriasis conditions for at least 3 months before screening (information obtained from medical chart or participant's physician, or directly from the participant)
* Participant has plaque psoriasis covering >= 1% but < 10% of his total BSA on Day 1
* For Group A: Participant has one psoriasis target lesion or individual lesions within the same anatomical region (excluding palms, soles, face, scalp, and genitals), with a target lesion severity score (TLSS) score of >= 6 on Day 1 allowing the collection of three microneedle device samples and one biopsy sample
* For Group B: Participant has one psoriasis target lesion or individual lesions within the same anatomical region (excluding palms, soles, face, scalp, and genitals), with a TLSS score of >= 6 on Day 1 allowing the collection of one microneedle device sample per visit (replicating the extraction on the same area at each visit) and one biopsy sample

Exclusion Criteria:

* Participant is a female who is breastfeeding, pregnant, or who is planning to become pregnant during the study
* Participant has evidence of erythrodermic, pustular, predominantly guttate psoriasis, or drug-induced psoriasis
* Participant has a history of skin disease or presence of skin condition that, in the opinion of the investigator, would interfere with the sample collection or interpretation
* Participant is known to have immune deficiency or is immunocompromised
* Participant has a history of cancer or lymphoproliferative disease within 5 years prior to Day 1. Participants with successfully treated nonmetastatic cutaneous squamous cell or basal cell carcinoma and/or localized carcinoma in situ of the cervix are not to be excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with mild chronic plaque psoriasis vulgaris, defined as having a body surface area (BSA) greater than or equal to (>=) 1 percent (%) and less than (<) 10% (excluding palms, soles, face, scalp, and genitals), will be included in this study.
Sampling Method: Probability Sample
Enrollment: 11 (Actual)
Dates: Start 2019-03-15 (Actual); Primary Completion 2019-11-25 (Actual); Study Completion 2019-12-06 (Actual)

PRIMARY OUTCOMES:
Measurement of Expression by RNA-sequencing (RNAseq) of Extracted RNA Using Punch Biopsy Method Versus Microneedle Device Sampling Method | Up to 28 days
  Measurement of expression by ribonucleic acid (RNA)-sequencing of extracted RNA by the frequently used punch biopsy method and the microneedle device will be performed to have a comparison between both the methods.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Innovaderm Research Inc., Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No